CLINICAL TRIAL: NCT04535999
Title: Phase IV Open Label Study of the Effects of Secukinumab on Nail Psoriasis and Non-Invasive Measures of Enthesitis
Brief Title: Open Label Study of the Effects of Secukinumab on Nail Psoriasis and Non-Invasive Measures of Enthesitis (Phase IV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 834149
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Intervention-Secukinumab
Masking Description: Open Label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Secukinumab
  Interventions: Drug: Secukinumab Auto-Injector

INTERVENTIONS:
Drug: Secukinumab Auto-Injector — 300 mg- Every 4 weeks after loading dose (Loading Dose-300 mg once weekly for 5 weeks)
  Other Names: Cosentyx

SUMMARY:
This study will be an open label study of secukinumab for the treatment of nail psoriasis. Secukinumab is an FDA-approved treatment for psoriasis. We will examine time to response and different methods of defining nail disease response.

DETAILED DESCRIPTION:
This study will be an open label study of secukinumab for the treatment of nail psoriasis. Secukinumab is an FDA-approved treatment for psoriasis. This is a single arm trial - all patients will receive the study drug. We will examine time to response and different methods of defining nail disease response.

ELIGIBILITY:
Inclusion Criteria:

* Active psoriatic nail disease defined as a Minimum 4 or more fingernails OR NAPSI>20
* Active skin psoriasis currently (no minimum PASI or BSA) or skin psoriasis in the past documented by a dermatologist
* Age 18-85

Exclusion Criteria:

* History of IL-17 inhibitor use (other therapies including TNF inhibitors or non- biologics DMARDS in the past are acceptable)
* Inflammatory bowel disease
* Metal implants or other concerns for use of MRI
* Active infection
* Patients may have a history of self-reported psoriatic arthritis but may not have active PsA at the time of screening.
* We will exclude patients with onychomyosis of the fingernails on clippings

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
NAPSI | Baseline to 24 Weeks
  Nail Psoriasis Severity Index (NAPSI): NAPSI is the most comprehensive nail assessment used in clinical trials. The fingernail is divided into four quadrants. For each quadrant, 1 point is assigned for a nail matrix abnormality and 1 point for a nail bed abnormality allowing for a total of 8 points per nail. 0-80 total points possible with a higher score corresponding to a worse outcome.

SECONDARY OUTCOMES:
PASI | Baseline to 24 Weeks
  Psoriasis Area Severity Index (PASI): Four assessments for each of four body areas (head, trunk, upper extremities, and lower extremities) are provided. The assessments are erythema, induration, and scale (each assessed as 0-4 using a standardized scale), and the number of palms/percentage of each area is categorized (0 = 0%, 1 = less than 10%, 2 = 10%-29%, 3 = 30%-40%, 4 = 50%-69%, 5 = 70%-89%, and 6 = 90%-100%). The scale is 0 to 72 with a higher score corresponding to a worse outcome.
Physician Global Assessment of Nail Disease | Baseline to 24 Weeks
  Physician Global Assessment of Nail Disease. Scale of 0-100 with higher score corresponding to a worse outcome.
DLQI | Baseline to 24 Weeks
  Dermatology Life Quality Index (DLQI):
  There are a total of 10 questions and each question is scored on a four-point Likert scale:
  Very much = 3 A lot = 2 A little = 1 Not at all = 0 Not relevant = 0 Question unanswered = 0
  The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ogdie-Beatty, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania, United States